CLINICAL TRIAL: NCT03943004
Title: A Phase I Study of DFP-14927 in Patients With Advanced Solid Tumors
Brief Title: Trial of DFP-14927 in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Delta-Fly Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D18-11161
Record Dates: First submitted 2019-04-25; First posted 2019-05-08 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor; Cancer
Keywords: advanced solid tumors; refractory or relapsed tumors
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DFP-14927 (Experimental): DFP-14927: weekly IV infusion, 28 day treatment cycle
  Interventions: Drug: DFP-14927

INTERVENTIONS:
Drug: DFP-14927 — DFP-14927 is a large 4-arm-PEGylated-DFP-10917 molecule. DFP-10917 is a nucleoside analog similar to deoxycytidine.

SUMMARY:
This is a Phase I, open-label, single-arm, dose escalation study of DFP-14927 intravenous infusion administered to patients with refractory or relapsed solid tumors.

DETAILED DESCRIPTION:
This study will determine the safety and efficacy of DFP-14927 in patients with refractory or relapsed advanced solid tumors. The study will be guided by a standard "3+3"dose escalation by observing the drug-related toxicities and dose-limiting toxicities following weekly IV infusion of DFP-14927 for each 28-day cycle (4 doses per cycle). In addition, the maximum-tolerated dose and recommended Phase II dose for DFP-14927 will be determined.

Furthermore, the study will determine the pharmacokinetics and bioavailability of DFP-14927 during the first cycle of treatment using the weekly dosing schedule.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically (or cytologically) confirmed diagnosis of solid tumor, refractory after standard therapy for the disease or for which conventional systemic therapy is not reliably effective or no effective therapy is available. Note: For expansion cohorts patients must have histologically (or cytologically) confirmed diagnosis of gastroesophageal cancer, pancreatic cancer, or cholangiocarcinoma that has relapsed or is refractory to standard therapy.
2. Aged ≥ 18 years.
3. ECOG Performance Status of 0 or 1.
4. Adequate clinical laboratory values defined as:

   1. absolute neutrophil count ≥ 1.5 x 10⁹/L
   2. platelets ≥ 100 x 10⁹/L
   3. hemoglobin ≥ 9.0 g/dL (transfusions permissible)
   4. plasma creatinine ≤ 1.5 x upper limit of normal (ULN) for the institution or calculated clearance ≥ 60 mL/min (Cockcroft-Gault formula)
   5. total bilirubin ≤ 1.5 x ULN
   6. alanine transaminase (ALT) and aspartate transaminase (AST) < 2.5 x ULN (<5 x ULN if documented hepatic metastases)
   7. prothrombin time (PT) ≤1.2 x ULN, partial thromboplastin time (PTT) ≤ 1.2 ULN, and international normalized ratio (INR) ≤ 1.5
5. Absence of uncontrolled intercurrent illnesses, including uncontrolled infections, cardiac conditions, uncontrolled diabetes mellitus, or other organ dysfunctions.
6. Patients may have measurable or non-measurable disease as defined by RECIST 1.1.
7. Signed Informed-consent prior to the start of any study specific procedures.
8. Women of child-bearing potential must have a negative serum or urine pregnancy test. Male and female patients must agree to use acceptable contraceptive methods for the duration of the study and for at least one month after the last drug administration.

Exclusion Criteria:

1. Patients will be excluded if they have received previous chemotherapy, immunotherapy, radiotherapy or any other investigational therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) or 5 half-lives for targeted therapies prior to this study entry.
2. Have not recovered from adverse events (must be Grade ≤1) due to agents administered more than 4 weeks earlier.
3. Have had any major bleeding episodes (variceal bleeds, hemorrhagic strokes, internal abdominal bleeds, etc.) within 6 months prior to starting study drug.
4. Known hypersensitivity to any study drug component (such as pegylated medications).
5. Extensive prior radiotherapy, more than 30% of bone marrow reserves, or prior bone marrow/stem cell transplantation.
6. Any concomitant condition that in the opinion of the investigator could compromise the objectives of this study and the patient's compliance.
7. Pregnant or lactating individuals.
8. Current malignancies of another type, with the exception of adequately treated in situ cervical cancer and basal cell skin cancer or other malignancies with no evidence of disease for 2 years or more.
9. Known history of HIV, HBV or HCV infection.
10. Documented or known bleeding disorder.
11. Requirement for anticoagulation treatment that increases INR or aPTT above the normal range (low dose DVT or line prophylaxis is allowed).
12. Clinically evident CNS metastases or leptomeningeal disease not controlled by prior surgery or radiotherapy; history of seizure disorder not controlled by anti-seizure medication at the time of enrollment. Patients with primary CNS malignancies are excluded.
13. Patients with a significant cardiovascular disease or condition, including:

    1. Myocardial infarction within 6 months of study entry
    2. NYHA Class III or IV heart failure
    3. Uncontrolled dysrhythmias or poorly controlled angina.
    4. History of serious ventricular arrhythmia (VT or VF, ≥ 3 beats in a row) and/or risk factors (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
    5. Baseline prolongation of QT/QTc interval (repeated demonstration of QTc ≥ 450 msec for men and 470 msec for women). QTc values up to 500 msec will be acceptable where patient's medical history, e.g. bundle branch block, is known to cause mild QTc prolongation and the condition is well controlled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) | From first dose (Day 1) up to 30 days after last dose
  The highest dose level at which less than one-third of at least 6 patients (i.e., 0 or 1 out of 6) experience a DLT
Recommended Phase II Dose (RP2D) | From first dose (Day 1) up to 30 days after last dose
  The maximum tolerated dose (MTD) of DFP-14927 at which the Phase II study will explore
Dose-Limiting Toxicity (DLT) | From first dose (Day 1) up to 30 days after last dose
  Determined through the frequency/severity of adverse events per CTCAE V5.0

SECONDARY OUTCOMES:
Determine objective response rate (CR or PR) in response to DFP-14927 study treatment | At pre-study and every 8 weeks through study completion, an average of 6 months
  Response to treatment will be assessed per RECIST 1.1
Duration of response | At pre-study and every 8 weeks through study completion, an average of 6 months
  Number of days from the time of initial response (CR or PR) to disease progression or death
PK parameters to be determined using area under the concentration curve (AUC) | Cycle 1 (each cycle is 28 days), Day 1: 0, 1, 2, 4, 8, 24, 48, and 96 hours post-dose; Day 8: 0,1, 2, 4, 8, 24, 48, and 96 hours post-dose and predose on Days 15, 22, and 29 (same as Day 1 of next Cycle)
  The concentration of DFP-14927 in blood plasma vs time
PK parameters to be determined using maximum drug concentration (Cmax) | Cycle 1 (each cycle is 28 days), Day 1: 0, 1, 2, 4, 8, 24, 48, and 96 hours post-dose; Day 8: 0,1, 2, 4, 8, 24, 48, and 96 hours post-dose and predose on Days 15, 22, and 29 (same as Day 1 of next Cycle)
  The maximum concentration of DFP-14927 in blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer Ajani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - UCLA Department of Medicine- Hematology/Oncology, Los Angeles, California
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No